CLINICAL TRIAL: NCT02721173
Title: Comparison of Safety and Efficacy of Tazarotene 0.1% Plus Clindamycin 1% Gel vs. Adapalene 0.1% Plus Clindamycin 1% Gel in the Treatment of Facial Acne Vulgaris: A Randomized Controlled Trial
Brief Title: Tazarotene Plus Clindamycin vs. Adapalene Plus Clindamycin in the Treatment of Facial Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Chandra Sekhar Sirka, Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM -NF/Derma/15/28
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Acne Vulgaris
Keywords: Tazarotene; Adapalene; Clindamycin
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene; Gels; Clindamycin; Adapalene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tazarotene group (Experimental): This group will receive tazarotene 0.1% gel plus clindamycin 1% gel for 4 weeks.
  Interventions: Drug: Tazarotene 0.1% gel plus clindamycin 1% gel
- Adapalene group (Active Comparator): This group will receive adapalene 0.1% gel plus clindamycin 1% gel for 4 weeks.
  Interventions: Drug: Adapalene 0.1% gel plus clindamycin 1% gel

INTERVENTIONS:
Drug: Tazarotene 0.1% gel plus clindamycin 1% gel — Medications will be advised to apply once daily in the evening after facial cleansing. Clindamycin will be applied first and tazarotene will be applied 5-10 minutes later.
  Arms: Tazarotene group
Drug: Adapalene 0.1% gel plus clindamycin 1% gel — Medications will be advised to apply once daily in the evening after facial cleansing. Clindamycin will be applied first and adapalene will be applied 5-10 minutes later.
  Arms: Adapalene group

SUMMARY:
The combination therapy of retinoid and clindamycin for acne is preferred because it targets multiple areas of acne pathogenesis that could not be accomplished with monotherapy, thereby improving outcome. Literature review reveals that till date there is no published comparative study assessing safety and efficacy of tazarotene plus clindamycin and adapalene plus clindamycin. So the present study has been designed to compare these two combination therapy in acne vulgaris.

DETAILED DESCRIPTION:
Acne vulgaris is one of the most common disorders treated by dermatologists. The pathogenesis of acne is multifactorial. Critical components include abnormal follicular keratinocyte desquamation leading to the formation of a follicular plug (microcomedo), increase of sebum production in pilosebaceous unit, colonization by Propionibacterium acnes, and inflammation. Topical retinoids, which target comedogenesis and have anti-inflammatory activity, are recommended as first-line therapy for both inflammatory and non-inflammatory acne. The adjunctive use of anti-acne agents like clindamycin by its complementary mechanism of action can help to enhance the efficacy of topical retinoid therapy still further.

Tazarotene is a synthetic retinoid and a prodrug that is converted by the skin to its active form, tazarotenic acid. The active form binds to retinoic acid receptors (RARs) and regulates gene transcription and helps to normalize the abnormal keratinization in the follicular infundibulum, this in turn changes the microenvironment of the follicle and thereby reduce the proliferation of Propionibacterium acnes. Adapalene is a synthetic naphthoic acid derivative with retinoid activity. Adapalene also acts through RARs and modulates cellular keratinization and inflammatory process. Clindamycin is bactericidal to Propionibacterium acnes. Due to the inhibition of P. acnes the free fatty acid levels in the pilosebaceous unit of skin is also reduced. Clindamycin phosphate applied topically penetrates to a very great extent to open comedones and thus produces a high percentage of sterile comedones.

The combination therapy of retinoid and clindamycin for acne is preferred because it targets multiple areas of acne pathogenesis that could not be accomplished with monotherapy, thereby improving outcome. Literature review reveals that till date there is no published comparative study assessing safety and efficacy of tazarotene plus clindamycin and adapalene plus clindamycin. So the present study has been designed to compare these two combination therapy in acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the diagnosis of facial acne vulgaris having comedones, papules, pustules (≤5), or nodules (≤2) or Investigator's static global assessment score ≤4
* Treatment naïve patients or patients who had not taken topical anti-acne medications in last 14 days, systemic antibiotics in last 30 days, oral retinoids in last 12 months

Exclusion Criteria:

* Very severe acne vulgaris (Investigator's static global assessment score >4)
* Any skin disorder that might interfere with the diagnosis or evaluation of acne vulgaris
* Known hypersensitivity to retinoids and clindamycin
* Any uncontrolled systemic disease or any cosmetic or surgical procedures complementary to the treatment of acne in the preceding 15 days
* Patients who were on oral contraceptive pills in last 12 weeks
* Pregnant and nursing women

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The number of facial acne lesions | Change from baseline over 4 weeks
  Total number of facial acne lesions (inflammatory and non-inflammatory) will be counted

SECONDARY OUTCOMES:
Severity of acne | Change from baseline over 4 weeks
  Severity of acne will be assessed by Acne global severity scale
Severity of acne | Change from baseline over 4 weeks
  Severity of acne will be assessed by Investigator's static global assessment (ISGA) score
Quality of life | Change from baseline over 4 weeks
  Quality of life will be assessed by Acne-specific quality of life questionnaire (Acne-QoL).

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, DM, Study Director — AIIMS, Bhubaneswar
Locations (1):
- AIIMS, Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Millikan LE. The rationale for using a topical retinoid for inflammatory acne. Am J Clin Dermatol. 2003;4(2):75-80. doi: 10.2165/00128071-200304020-00001. PMID 12553848
- [Result] Jeremy AH, Holland DB, Roberts SG, Thomson KF, Cunliffe WJ. Inflammatory events are involved in acne lesion initiation. J Invest Dermatol. 2003 Jul;121(1):20-7. doi: 10.1046/j.1523-1747.2003.12321.x. PMID 12839559
- [Result] Do TT, Zarkhin S, Orringer JS, Nemeth S, Hamilton T, Sachs D, Voorhees JJ, Kang S. Computer-assisted alignment and tracking of acne lesions indicate that most inflammatory lesions arise from comedones and de novo. J Am Acad Dermatol. 2008 Apr;58(4):603-8. doi: 10.1016/j.jaad.2007.12.024. Epub 2008 Feb 4. PMID 18249468
- [Result] Talpur R, Cox K, Duvic M. Efficacy and safety of topical tazarotene: a review. Expert Opin Drug Metab Toxicol. 2009 Feb;5(2):195-210. doi: 10.1517/17425250902721250. PMID 20213916
- [Result] Thiboutot D, Gollnick H, Bettoli V, Dreno B, Kang S, Leyden JJ, Shalita AR, Lozada VT, Berson D, Finlay A, Goh CL, Herane MI, Kaminsky A, Kubba R, Layton A, Miyachi Y, Perez M, Martin JP, Ramos-E-Silva M, See JA, Shear N, Wolf J Jr; Global Alliance to Improve Outcomes in Acne. New insights into the management of acne: an update from the Global Alliance to Improve Outcomes in Acne group. J Am Acad Dermatol. 2009 May;60(5 Suppl):S1-50. doi: 10.1016/j.jaad.2009.01.019. PMID 19376456
- [Result] Draelos ZD, Tanghetti EA; Tazarotene Combination Leads to Efficacious Acne Results (CLEAR) Trial Study Group. Optimizing the use of tazarotene for the treatment of facial acne vulgaris through combination therapy. Cutis. 2002 Feb;69(2 Suppl):20-9. PMID 12095065
- [Result] Piskin S, Uzunali E. A review of the use of adapalene for the treatment of acne vulgaris. Ther Clin Risk Manag. 2007 Aug;3(4):621-4. PMID 18472984
- [Result] Feldman SR, Werner CP, Alio Saenz AB. The efficacy and tolerability of tazarotene foam, 0.1%, in the treatment of acne vulgaris in 2 multicenter, randomized, vehicle-controlled, double-blind studies. J Drugs Dermatol. 2013 Apr;12(4):438-46. PMID 23652892
- [Result] Adityan B, Kumari R, Thappa DM. Scoring systems in acne vulgaris. Indian J Dermatol Venereol Leprol. 2009 May-Jun;75(3):323-6. doi: 10.4103/0378-6323.51258. No abstract available. PMID 19439902
- [Result] Martin AR, Lookingbill DP, Botek A, Light J, Thiboutot D, Girman CJ. Health-related quality of life among patients with facial acne -- assessment of a new acne-specific questionnaire. Clin Exp Dermatol. 2001 Jul;26(5):380-5. doi: 10.1046/j.1365-2230.2001.00839.x. PMID 11488820
- [Derived] Maiti R, Sirka CS, Ashique Rahman MA, Srinivasan A, Parida S, Hota D. Efficacy and Safety of Tazarotene 0.1% Plus Clindamycin 1% Gel Versus Adapalene 0.1% Plus Clindamycin 1% Gel in Facial Acne Vulgaris: A Randomized, Controlled Clinical Trial. Clin Drug Investig. 2017 Nov;37(11):1083-1091. doi: 10.1007/s40261-017-0568-2. PMID 28913735